CLINICAL TRIAL: NCT04794777
Title: A Randomized Trial Comparing Conventional "Salvage" Radiotherapy and Individualized 68Ga-PSMA-11 or 18F-PSMA-1007 PET/CT Targeted Treatment in Patients With Biochemical Recurrence After Prostate Cancer Surgery
Brief Title: Comparing "Salvage" Radiotherapy and Individualized PSMA PET/CT Targeted Treatment in With Relapsing Prostate Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stefan Carlsson (Other)
Responsible Party: Sponsor-Investigator, Stefan Carlsson, Principal Investigator, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSMA recidiv
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
Keywords: PSMA PET/CT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm (Experimental): Individualised therapy based on results of the PSMA PET/CT.
  Interventions: Combination Product: Individualised therapy
- Control arm (Active Comparator): Standard salvage therapy. Results of PSMA PET/CT blinded.
  Interventions: Radiation: Standard salvage therapy

INTERVENTIONS:
Combination Product: Individualised therapy — Group I - No uptake: treated with conventional SRT against the prostate bed. Group II -Uptake only in the prostate bed: will receive intensity modulated RT (IMRT) including Volumetric Modulated Arc Therapy (VMAT) for prostate bed with simultaneous-integrated boost (SIB) to the PET positive uptake in the prostate bed.
  Group III - Uptake in the prostate bed and involvement of regional lymph nodes in the pelvis: will be treated as Group II plus VMAT for the pelvic lymph nodes with SIB to the PET positive lymph nodes or pelvic lymph nodes salvage lymph node dissection (SLND).
  Group IV - Uptake in regional lymph nodes only: will be treated with VMAT for the pelvic lymph nodes with SIB to the PET positive lymph nodes or pelvic lymph nodes SLND.
  Group V - Uptake in extra-pelvic lymph nodes or bone metastasis: systemic treatment instead of surgery or radiation. Local treatment with surgery or radiation is acceptable if curative intention.
  Arms: Experimental arm
Radiation: Standard salvage therapy — Standard salvage radiotherapy
  Arms: Control arm

SUMMARY:
Less than 50% of patients receiving salvage radiation therapy (SRT) to the pelvis as treatment for prostate cancer relapsing after surgery will achieve undetectable Prostate Specific Antigen (PSA) levels. Despite SRT, two-thirds of patients will again develop elevated PSA, 20% will have distant metastases, and 10% will die from prostate cancer within 10 years. The reason for this is probably preexisting distant metastasis and lymph node metastasises which need to better targeted directly. Additionally , there are well known permanent side effects to SRT.

Standard imaging techniques have poor sensitivity detecting recurrence when PSA is below 1.0 ng/ml. The surface protein Prostate-specific membrane antigen (PSMA) is overexpressed on prostate cancer cells and 68Gallium (68Ga)- and 18Fluorine (18F)-targeted radioligands have been developed. PSMA PET/CT is used increasingly but there is limited data of its impact.

In this study patients with biochemical relapse of prostate cancer after surgery are randomised to the control or experimental group (1:2) and undergo a PSMA PET/CT scan. The experimental group receives individualised therapy based on the result of the PET/CT. The control group receives standard salvage therapy and the result of the PET/CT is blinded. The patients are followed-up with PSA test and quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously treated for prostate cancer with radical prostatectomy and now having a biochemical recurrence (BCR) defined as: PSA >0.2 <2.0 ng/mL, and increasing measured twice.
* Multidisciplinary conference (MDK) decision to offer the patient SRT
* Signed Informed Consent

Exclusion Criteria:

* Patients previously treated for prostate cancer with biochemical recurrence
* Previous treatment with androgen deprivation therapy (ADT) after surgery
* Previous pelvic radiotherapy
* Patients with positive lymph nodes at surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2018-10-30 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Primary PSA progression free survival | Throughout the study, approximately 10 years.
  Number of patients with progress defined by Prostate-Specific Antigen (PSA) measurement

SECONDARY OUTCOMES:
Time to metastasis | At 5, 7 and 10 years
  Time to documented metastasis of prostate cancer
Prostate cancer specific survival | At 5, 7 and 10 years
  Time to prostate cancer specific death
Time to secondary treatment | At 5, 7 and 10 years
  Time to need for secondary treatment for prostate cancer
Differences in quality of life recorded using Patient Reported Outcome Measure (PROM) | Baseline, 6, 12, 36 and 60 months after completed treatment.
  A modified version of the PSMA questionnaire developed by the National Prostate Cancer Register. Scale from 1 to 5 were 1 is very good and 5 is very bad.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Carlsson, Principal Investigator — Karolinska University Hospital
Locations (5):
- Sweden (5):
  - Sahlgrenska University Hospital, Gothenburg, Göteborg
  - Södersjukhuset, Stockholm, Stockholm County
  - Karolinska University Hospital, Stockholm, Stockholm County
  - Norrland's University Hospital, Umeå
  - Örebro University Hospital, Örebro, Örebro County

IPD SHARING:
Plan to Share IPD: No